CLINICAL TRIAL: NCT01480986
Title: a Prospective Study on the Efficacy and Safety Using Sequential Therapy of Irinotecan Combined With Cisplatin (IP)and Octretide Lar in the First Line Treatment of Metastatic or Inoperable Gastrointestinal Poorly Differentiated Neuroendocrine Carcinoma: the IPO-NEC Trial
Brief Title: IPO-NEC Trial:Study on the Efficacy and Safety Using Sequential IP Therapy and Oct Lar in the Treatment of Advanced GI NEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Head of GI Cancer department, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJT-NEC-001
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Progression Free Survival of the Treatment
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): This is a single arm trial. The patient will enter phase one and will continue to phase two once the disease progresses in phase one or the phase one has been completed.
  Interventions: Drug: Irinotecan combined with cisplatin, octreotide lar

INTERVENTIONS:
Drug: Irinotecan combined with cisplatin, octreotide lar — Phase 1 irinotecan 180mg/m^2，ivgtt，90min，D1 Cisplatin 50 mg/m^2，ivgtt，120min，D1（with hydration） Phase 2 Octreotide 0.1mg，ih，q8h，D1-14 Octreotide lar 20mg，deep i.m，D8，

SUMMARY:
This is a prospective, single-armed, open label study on the efficacy and safety of sequential IP therapy(Irinotecan plus cisplatin) and octreotide lar in the treatment of GI poorly diffrentiated Neuroendocrine carcinoma. Patient with written consents will enter the phase one step of the trial, receiving IP therpy. Once the IP therapy has been finished without disease progression or progression occurs during the treatment, the patient will enter the phase two step of the trial, receiving octreotide treatment. The primary endpoint is progression free survival in the two steps respectively and secondary endpoint is disease control rate, overall survival and safety

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent
* Male or female patients >=18 years old
* Histologically or cytologically confirmed poorly differentiated neuroendocrine carcinoma originating from the GI tract. The grade of the disease is grade 2 or grade 3
* No previous treatment is allowed including chemotherapy, radiotherapy,immunotherapy or others. In case the patient received adjuvant therapy after surgery, enrollment is allowed if the adjuvant therapy doesn't contain cisplatin or irinotican and at the same time, the last day of chemotherapy is ≥180 days before screening.
* Target lesion more than 1cm in diameter by enhanced CT or MRI 21 days before enrollment
* The laboratory parameter meets the following criteria 7 days before enrollment
* Hemoglobin ≥90g/L
* Absolute neutrophil count≥1.5×10^9/L, platelets 100×10^9/L；
* ALT and AST≤2.5 ULN(in case of the patients with liver metastasis,ALT and AST≤5.0 ULN)
* ALP ≤2.5 ULN (in case of the patients with liver metastasis,≤5.0 ULN)
* Total Serum bilirubin ≤1.5 ULN
* Serum creatinine ≤1.0 ULN
* KPS ≥70
* Estimated survival ≥90 days
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days of enrollment and must be willing to use adequate methods of contraception during the study and for 30 days after last study durg administration.

Exclusion Criteria:

* Known sensitivity to 5-HT3 antagonist and hypersensitivity to the other treatment agents including irinotecan, cisplatin and octreotide lar
* Any participation in trials simultaneously or 4 weeks before screening.
* Undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such surgery.
* Uncontrolled severe diarrhea
* Unconrolled active infection (fever ≥38 degrees due to infection)
* severe hepatopathy including active hepatitis and hepatic cirrhosis, renal dysfunction, severe pulmonary diseases including interstitial pneumonia, pulmonary fibrosis and severe pulmonary emphysema, uncontrolled diabetes, hypertension and other chronic systematic diseases.
* Chronic treatment with steroids.(In case of the patients with short-term use of steroids, the enrollment is permitted if the administration is stopped 2 weeks before screening.)
* confirmed or suspected CNS metastasis
* the history of peripheral nervous system impairment, obvious mental disorder or CNS impairment
* clinically significant heart disease, including congestive heart failure, symptomatic coronal heart disease, arrythmia uncontrolled by medication and acute myocardial infarction or cardiac insufficiency within 6 months before screening
* pregnant women or women in lactation period
* Fertile male or women of child-bearing potential refuse to take highly effective methods of birth control
* Incidence of other second primary malignant tumors, except for cured basal cell carcinoma and cervical carcinoma in situ.
* patients of legal incapacity or who have the potential of influence the whole trial due to medical or ethic reasons.
* Other patients who are not eligible to the trial under investigators' discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival for Irinotecan plus cisplatin and octreotide | 2 years
  The primary objective is to investigate the overall progression free suvival for irinotecan plus cisplatin and octretide. The respective PFS of the two treatment steps will also be investigated. The result will be compared with the history treatment outcomes for patients of poorly differentiated neuroendocrine carcinoma.

SECONDARY OUTCOMES:
Disease control rate | 2 years
  The second objective includes the disease control rate of irinotecan plus cisplatin and octretide theray.
Overall survival | 3 years
  The secondary objective includes the investigation of the overall survival for the patients receiving the sequential treatment of irinotecan plus cisplatin and octretide.
Safety | 3 years
  The secondary objective also includes the investigation on the safety profiles of the two interventions, irinotecan plus cisplatin treatment and octretide. The safety profile will be described using incidence of AEs and SAEs, using CTCAE criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tumor Hospital, Beijing, Beijing Municipality, China